CLINICAL TRIAL: NCT00534118
Title: Cellular Infusions in Patients With Recurrent or Persistent Hematologic Malignancies After Allogeneic Stem Cell Transplant
Brief Title: Donor Lymphocyte Infusion in Treating Patients With Recurrent or Persistent Hematologic Cancer After Donor Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564827; RPCI-I-00703
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; childhood chronic myelogenous leukemia; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; de novo myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; cutaneous B-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Hodgkin Disease; Recurrence; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infusion (Experimental): Patients receive up to four donor lymphocyte infusions at least 1 month apart in the absence of disease progression, unacceptable toxicity, or uncontrolled graft-versus-host disease
  Interventions: Biological: donor lymphocytes

INTERVENTIONS:
Biological: donor lymphocytes — Given IV

SUMMARY:
RATIONALE: Giving an infusion of donor lymphocytes may be able to kill cancer cells in patients with hematologic cancer that has come back after a donor stem cell transplant.

PURPOSE: This clinical trial is studying how well donor lymphocyte infusion works in treating patients with recurrent or persistent hematologic cancer after donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if the complete response rate exceeds 10% in patients with recurrent or persistent hematologic malignancies treated with donor lymphocyte infusion.

Secondary

* Estimate the complete response rate in these patients.
* Assess the toxicity of donor lymphocyte infusion in these patients.

OUTLINE: Patients receive up to four donor lymphocyte infusions at least 1 month apart in the absence of disease progression, unacceptable toxicity, or uncontrolled graft-versus-host disease.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Has undergone allogeneic stem cell transplantation (ASCT) for hematologic malignancy at least 30 days ago

  * No failure to engraft following transplant
  * No active acute or chronic graft-versus-host disease (GVHD)

    * Minimal GVHD allowed
* Persistent or relapsed disease after ASCT, including 1 of the following:

  * Chronic myelogenous leukemia (CML), meeting any of the following criteria:

    * Molecular relapse (may be treated with imatinib mesylate after transplant), as defined by any of the following:

      * ASCT was non-T-cell depleted, a negative bcr/abl was documented by PCR post-transplant, and bcr/abl is now detectable by 2 consecutive PCR determinations > 30 days apart
      * ASCT was non-T-cell depleted and bcr/abl is detectable by PCR at any time after day 180 post-transplant
    * Cytogenetic relapse after 3-6 months of imatinib mesylate
    * Relapsed chronic phase, accelerated phase, or blastic phase CML after 3-6 months of imatinib mesylate

      * Must currently be in chronic phase or accelerated phase CML only
      * Patients with blastic phase CML must attain a second chronic phase
  * Acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes, meeting any of the following criteria:

    * Molecular relapse, as evidenced by < 5% blasts in the bone marrow and the patient's leukemia-specific molecular abnormality detectable by PCR
    * Cytogenetic relapse, as evidenced by < 5% blasts in the bone marrow and the patient's leukemia-specific chromosome abnormality detectable by standard cytogenetics at any time after day 60 post-transplant
    * Hematologic relapse, as evidenced by > 20% blasts in bone marrow or soft tissue recurrence

      * Must be treated with chemotherapy after transplant, but before study donor lymphocyte infusion (DLI)
  * Multiple myeloma

    * Relapsed disease or recurrence of M-protein after thalidomide or other salvage treatment

      * Prior post-transplant documentation of disappearance of M-protein by immunofixation
    * Residual or progressive disease
    * Rising M-protein level at any time post-transplant (measured at 3-month intervals)
    * Original M-protein detectable at 6 months post-transplant
    * Immune protein electrophoresis (IPEP) is required to show that M-component is the same on day 60 post-transplant as pre-transplant
    * Residual (> 5%) plasma cells in bone marrow
  * Relapsed non-Hodgkin lymphoma or Hodgkin lymphoma

    * Relapse or progression of disease must be evidenced within 3 months prior to donor lymphocyte infusion by physical exam, radiographic studies, or molecular studies

      * Tumor should be re-biopsied to determine histology
    * If Epstein-Barr virus (EBV) lymphoma is suspected, peripheral blood must be assayed for EBV genome (i.e., EBV DNA testing by PCR) within the past 30 days
  * EBV infection with associated pancytopenia

    * Persistent or refractory pancytopenia with EBV genome detected by PCR in the peripheral blood

      * Refractory pancytopenia is defined as pancytopenia that is poorly responsive to growth factors and/or transfusions
  * EBV lymphoproliferative disorder

    * Clonal lymphadenopathy that is refractory to standard therapy with acyclovir and immunoglobulin (DLI may be given with rituximab)
* Not a candidate for repeat ASCT

  * Chimerism status is not required for determining eligibility for DLI
* Patients eligible for allogeneic ASCT, but for whom DLI is offered as the first option, should have full donor chimerism at relapse or after therapy for relapsed disease
* Patients with relapsed underlying disease after transplant who achieved remission after chemotherapy are allowed
* No CNS recurrence that is not cleared by standard chemotherapy

  * CNS remission status must be maintained for 2 weeks
* Original hematopoietic progenitor stem cell donor must be available for cell donation

  * No syngeneic donors

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 8 weeks
* Creatinine < 3 mg/dL
* ABO/Rh and CMV IgG/IgM status known
* No HIV1 and HIV2 antibody
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months (males) or 6 months (females) after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple DLI: Accruals where the patient received 2-4 donor lymphocyte infusions Arm includes total number of infusions
- Single DLI: accruals where the patient received only one donor lymphocyte infusion
Period: Overall Study
Arm/Group | Multiple DLI | Single DLI
Started | 17 | 22
Completed | 17 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants can be accrued more than once; Accruals are based on the number of times the participant had a treatment (DLI) cycle that was evaluable (ie. >8 weeks between infusions per the protocol). DLIs which were given <8 weeks apart counted as one accrual.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple DLI | Single DLI | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 45 [16 to 66] | 53.5 [9 to 68] | 51 [9 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27
Disease [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 8 | 9 | 17
  Myelodysplastic Syndrome | 2 | 0 | 2
  Non Hodgkin Leukemia | 2 | 1 | 3
  Acute Lymphoblastic Leukemia | 1 | 0 | 1
  Chronic Myeloid Leukemia | 1 | 1 | 2
  Hodgkin Lymphoma | 1 | 0 | 1
  Prolymphocytic Leukemia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: continued or induced complete remission after DLI
Time Frame: 100 days post DLI
Population: Each accrual is evaluable independently, some patients in both the Multiple and Single DLI are accrued more than once; total unique patients in multiple DLI is 15 and in single DLI is 12
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple DLI | Single DLI
Number analyzed (Participants) | 17 | 22
Participants | 8 | 6

2. Primary Outcome: Duration of Complete Response in Months (Maximum 12)
Description: For participants who achieve a complete remission after DLI, the duration of time until 1) relapse or 2) death in remission or 3) subsequent DLI or 4) last followup (at 1 year after DLI)
Time Frame: 1 year post DLI
Population: Accruals which achieved a continued or induced complete remission at Day +100 after DLI, patients are censored at death in remission or at time of subsequent DLI
Measure: Median (Full Range); unit: months
Groups:
- Multiple DLI - Complete Responders; Single DLI - Complete Responders: Duration of time patients who achieved a complete remission by day +100 after DLI maintained that remission
Arm/Group | Multiple DLI - Complete Responders | Single DLI - Complete Responders
Number analyzed (Participants) | 8 | 6
months | 10.1 [1.7 to 12] | 9 [1.0 to 12]

3. Secondary Outcome: Acute Graft-versus-host Disease
Description: development of grade III-IV acute graft-versus-host disease (GVHD) per Glucksberg criteria
Time Frame: 100 days post DLI
Population: Each accrual is evaluable for acute GVHD grade III-IV
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple DLI | Single DLI
Number analyzed (Participants) | 17 | 22
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: All cause mortality includes individual participants who experienced death due to any cause before 3 years after first DLI and is the only SAE/AE captured per protocol
Description: All cause mortality includes individual participants who experienced death due to any cause before 3 years after first DLI
Arm/Group | Multiple DLI | Single DLI
All-Cause Mortality (participants affected / at risk) | 10/15 | 7/12
Serious Adverse Events (participants affected / at risk) | 10/15 | 7/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple DLI (N=15) | Single DLI (N=12)
All cause mortality by 3 years after first DLI (General disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT00534118/Prot_SAP_000.pdf